CLINICAL TRIAL: NCT01643473
Title: Tailored Approaches to Improve Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: s14-00414
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Hypertension
Keywords: Hypertension; Latinos; Medication Adherence; Blood Pressure Control; Patient-centered; Black
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control (Active Comparator): Health education videos on topics unrelated to medication adherence, hypertension or type 2 diabetes
  Interventions: Other: Attention Control
- Tailored Adherence Intervention (Experimental): Tablet-based tailored adherence intervention matched to patients' most salient adherence barriers
  Interventions: Behavioral: Adherence Intervention

INTERVENTIONS:
Behavioral: Adherence Intervention — Patients randomized to the TAI group will complete a tailoring survey at the baseline visit to identify the most salient adherence barriers to the individual, which will be used to create an individualized adherence profile. Following completion of the tailoring survey, patients will collaborate with the RA to identify the most suitable mix of intervention strategies for improving medication adherence (i.e., reminder aids, motivational interviewing, case management) that are matched to the barriers outlined on patients' individualized adherence profiles.
  Arms: Tailored Adherence Intervention
Other: Attention Control — Health education videos on topics unrelated to medication adherence, hypertension or type 2 diabetes
  Arms: Attention Control

SUMMARY:
The purpose of this study is to to culturally tailor a technology-based individualized adherence intervention for Black and Latino patients with uncontrolled HTN or T2DM, who are non-adherent to their medications, and determine its acceptability.

DETAILED DESCRIPTION:
Using a randomized controlled trial design, this study will compare the efficacy of a tailored adherence intervention (TAI) to a single patient education (PE) session, on medication adherence among 40 high-risk Black and Latino patients with uncontrolled hypertension (HTN) who are non-adherent to their prescribed antihypertensive medications. Patients randomized to the PE group will receive a single tablet delivered patient education session at the baseline visit. Patients randomized to the TAI group will complete a tailoring survey at the baseline visit to identify the most salient adherence barriers to the individual, which will be used to create an individualized adherence profile. Following completion of the tailoring survey, patients will collaborate with the RA to identify the most suitable mix of intervention strategies for improving medication adherence (i.e., reminder aids, motivational interviewing, case management) that are matched to the barriers outlined on patients' individualized adherence profiles.

ELIGIBILITY:
Inclusion Criteria:

* Have uncontrolled hypertension defined as BP>140/90 mmHg on at least two consecutive visits in the past year (or BP>130/80 mmHg for those with diabetes or kidney disease) and Framingham Risk Scores (FRS) >20% (or at least one CVD risk factor including hyperlipidemia or diabetes);
* Have been prescribed at least one antihypertensive or oral anti-diabetic medication;
* Self-identify as Latino or African American/Black
* Be > 18 years of age

Exclusion Criteria:

* Refuse or are unable to provide informed consent;
* Currently participate in another hypertension study; or 2 diabetes study
* Have significant psychiatric comorbidity
* Plan to discontinue care at the clinic within the next 3 months

Vulnerable populations including adults unable to provide informed consent, pregnant women, and prisoners will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2018-02-20 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Schoenthaler, EdD, Principal Investigator — NYU Langone Health
Locations (1):
- Union Health Center, New York, New York, United States

REFERENCES:
- [Derived] Schoenthaler A, Leon M, Butler M, Steinhaeuser K, Wardzinski W. Development and Evaluation of a Tailored Mobile Health Intervention to Improve Medication Adherence in Black Patients With Uncontrolled Hypertension and Type 2 Diabetes: Pilot Randomized Feasibility Trial. JMIR Mhealth Uhealth. 2020 Sep 23;8(9):e17135. doi: 10.2196/17135. PMID 32965230
- [Derived] Schoenthaler A, De La Calle F, Barrios-Barrios M, Garcia A, Pitaro M, Lum A, Rosal M. A practice-based randomized controlled trial to improve medication adherence among Latinos with hypertension: study protocol for a randomized controlled trial. Trials. 2015 Jul 2;16:290. doi: 10.1186/s13063-015-0815-x. PMID 26134837

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Attention Control | Tailored Adherence Intervention
Started | 21 | 21
Completed | 20 | 21
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control | Tailored Adherence Intervention | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (11.3) | 59.7 (10.7) | 57.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 19 | 39
  White | 0 | 0 | 0
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Educational Status [Count of Participants; unit: Participants]
  Less than High School | 3 | 2 | 5
  High School Degree | 10 | 13 | 23
  Some College and above | 8 | 6 | 14
Unemployed [Count of Participants; unit: Participants] | 9 | 20 | 29
Annual income less than $40,000 [Count of Participants; unit: Participants] | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Retaining Study Participants Through the 3 Month Trial
Description: Feasibility is assessed as the absolute number of patients that are retained in the study once they are consented and enrolled at baseline.
Time Frame: 3 months
Population: The number of participants that were retained in the study from baseline to 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control | Tailored Adherence Intervention
Number analyzed (Participants) | 20 | 21
Participants | 20 | 21

2. Secondary Outcome: Change From Baseline in Mean Systolic and Diastolic Blood Pressure at 3 Months
Description: Change in mean systolic and diastolic blood pressure readings from baseline to 3 months. Systolic and diastolic blood pressure are measured in mmHg using a validated automated blood pressure monitor. The average of three readings was used as the blood pressure measurements for the baseline and 3 month study visit.
Time Frame: baseline and 3 months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Attention Control | Tailored Adherence Intervention
Number analyzed (Participants) | 20 | 21
mmHg
  Systolic blood pressure | -6.1 (3.9) | -7.2 (3.7)
  Diastolic blood pressure | -1.9 (2.3) | -3.5 (2.0)

3. Secondary Outcome: Change From Baseline in HbA1c at 3 Months
Description: Change in HbA1c from baseline to 3 months using a validated point-of-care device (Afinion AS100 Analyzer) at baseline and 3 months.
Time Frame: baseline and 3 months
Measure: Mean (Standard Error); unit: percentage of A1c
Arm/Group | Attention Control | Tailored Adherence Intervention
Number analyzed (Participants) | 20 | 21
percentage of A1c | 0.6 (0.49) | -0.5 (0.30)

4. Secondary Outcome: Change From Baseline in Self-reported Medication Adherence at 3 Months
Description: Medication adherence will be assessed by self-report using the validated 8-item Morisky Medication Adherence Scale. Scores range from 0-8, with higher scores indicative of better medication adherence.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Attention Control | Tailored Adherence Intervention
Number analyzed (Participants) | 20 | 21
score on a scale | 1.8 (0.49) | 1.3 (0.48)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Attention Control | Tailored Adherence Intervention
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT01643473/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT01643473/SAP_001.pdf